CLINICAL TRIAL: NCT01370096
Title: Vasopressin and Inhaled Prostacyclin in Pediatric Pulmonary Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty with patient recruitment
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Lindsay Ryerson, Assistant professor, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-LR-001
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Epoprostenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Vasopressin infusion — An intravenous infusion of vasopressin will be started at an initial rate of 0.0002U/Kg/min via the side arm of the central venous sheath. The infusion will be titrated up by 0.0001U/kg/min every minute until there has been a 20% increase in invasive mean arterial blood pressure (maximum infusion 0.002U/kg/min) and then the infusion may be titrated to maintain this blood pressure.
Drug: Vasopressin infusion and epoprostenol inhalation — An intravenous infusion of vasopressin will be started at an initial rate of 0.0002U/Kg/min via the side arm of the central venous sheath. The infusion will be titrated up by 0.0001U/kg/min every minute until there has been a 20% increase in invasive mean arterial blood pressure (maximum infusion 0.002U/kg/min) and then the infusion may be titrated to maintain this blood pressure. If the target 20% increase in SBP is not achieved with vasopressin titration, the infusion will remain at 0.002U/kg/min. After a period of ten minutes of drug exposure to allow for patient equilibration, subjects will receive nebulized prostacyclin at a dose of 50ng/kg/min for 15 minutes via Aeroneb into the endotracheal tube.
  Other Names: Flolan

SUMMARY:
To diagnose pulmonary hypertension, children have a cardiac catheterization to check the blood pressure in their lungs. Children with pulmonary hypertension have high blood pressure in their lungs. The right ventricle of the heart has to do more work to pump against this higher pressure. The investigators do not know the best medicine(s) to help children with pulmonary hypertension when their right ventricles fail. The purpose of the study is to look at the effects of two different medicines on the blood pressure in the lungs of a child with pulmonary hypertension. The investigators hope to then be able to choose the best medicine for children with pulmonary hypertension and right ventricular failure.

The first medicine is called vasopressin. It is a hormone that your body makes on its own. The investigators will be giving it through an intravenous infusion. The investigators think that vasopressin works differently in different parts of your body. The investigators are looking to see the different effects that vasopressin has in the lungs compared to the rest of the body.

The second medicine is called prostacyclin and is something that your body also makes by itself. Prostacyclin, given via an intravenous infusion, is a treatment for pulmonary hypertension as it decreases pressure in the blood vessels. In the catheterization laboratory, patients breathe in this medicine to measure specific changes in the blood pressure in their lungs.

DETAILED DESCRIPTION:
Background:

Pulmonary hypertension (PH) is a rare, but devastating disease that affects both adult and pediatric patients. Mortality is high with 84% survival at one year and 50% survival at five years in adult populations despite treatment. The cause of death is typically either from right ventricular failure or sudden cardiac death, likely secondary to a pulmonary hypertensive crisis. The resuscitation of patients with PH after cardiac arrest is extremely difficult. The use of epinephrine, a pulmonary vasoconstrictor, during resuscitation may impair filling of the left ventricle. The ideal resuscitation drug(s) would dilate the pulmonary vascular bed to help fill the left ventricle while constricting the systemic vascular bed to maintain coronary perfusion.

Objectives:

The assessment of pulmonary vascular reactivity is critical to the clinical management of patients with pulmonary hypertension (PH). The goals of this pilot study include determination of the hemodynamic effects of low dose vasopressin infusion and the effects of a combination of low dose vasopressin infusion and inhaled prostacyclin in a population of pediatric patients with PH.

Methods:

The investigators propose a prospective, pilot study to examine the acute hemodynamic effects of low dose vasopressin infusion and the combination of low dose vasopressin infusion and inhaled prostacyclin in pediatric pulmonary hypertension patients. The investigators anticipate recruiting 10 pediatric patients with pulmonary hypertension over the course of one year.

Study Protocol:

The study will be performed in the cardiac catheterization laboratory. All subjects will be intubated and mechanically ventilated for the study as per laboratory protocol. Sedation and anesthesia will be performed at the discretion of the pediatric anesthesiologist to provide a consistent anesthetic during the period of hemodynamic study. Arterial and venous access will be obtained via the femoral approach by standard techniques. Right and left catheterization will be performed to record hemodynamic measurements at baseline and after pulmonary vasoreactivity testing with oxygen and nitric oxide as per usual. Catheterization data to be collected includes right atrial pressure, systolic, diastolic and mean pulmonary artery pressure, pulmonary capillary wedge pressure, systemic arterial pressure, cardiac index, pulmonary vascular resistance (PVR) index, systemic vascular resistance (SVR) index and PVR/SVR ratio. After a period of time to allow for nitric oxide washout, acute vasoreactivity testing to assess the hemodynamic response to low dose vasopressin infusion followed by the combination of low dose vasopressin infusion and inhaled PGI2 will be performed.

ELIGIBILITY:
Inclusion Criteria:

All pediatric patients with pulmonary hypertension defined as a mean pulmonary artery pressure ≥ 25mmHg undergoing diagnostic cardiac catheterization for clinical purposes are potential subjects. Subjects must have preserved left ventricular function (ejection fraction ≥ 40 %). Subjects must have parental consent for enrollment.

Exclusion Criteria:

1. Any patient with left ventricular dysfunction (EF < 40%).
2. Any patient with known pulmonary veno-occlusive disease

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2012-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
PVR/SVR indexed ratio | Within 15 minutes of intervention
  Cardiac cath data

CONTACTS AND LOCATIONS:
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No